CLINICAL TRIAL: NCT01438814
Title: A Randomised, Double-blind, Double-dummy, Active-comparator Controlled Study Investigating the Efficacy and Safety of Linagliptin Co-administered With Metformin QD at Evening Time Versus Metformin BID Over 14 Weeks in Treatment Naive Patients With Type 2 Diabetes Mellitus and Insufficient Glycaemic Control
Brief Title: Linagliptin in Combination With Metformin in Treatment Naive Patients With Type 2 Diabetes Mellitus and Insufficient Glycaemic Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.60; 2011-002276-16 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-09-21; First posted 2011-09-22 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Linagliptin

ARMS (2):
- linagliptin + metformin (Experimental): patients to receive linagliptin +metformin QD
  Interventions: Drug: metformin; Drug: linagliptin
- metformin (Active Comparator): patients to receive metformin BID
  Interventions: Drug: metformin placebo; Drug: linagliptin placebo; Drug: metformin

INTERVENTIONS:
Drug: metformin placebo — metformin placebo tablets 500mg
  Arms: metformin
Drug: linagliptin placebo — linagliptin placebo tablets 5mg
  Arms: metformin
Drug: metformin — metformin tablets 500mg
  Arms: metformin
Drug: metformin — metformin tablets 500 mg
  Arms: linagliptin + metformin
Drug: linagliptin — linagliptin tablets 5mg
  Arms: linagliptin + metformin

SUMMARY:
The aim of this study is to investigate the impact of the combination therapy of linagliptin and metformin at submaximal doses in reduction of Glycosylated haemoglobin (HbA1c) and metformin pre-specified gastro-intestinal (GI) side effects in treatment naive patients of with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of Type 2 diabetes mellitus (T2DM) prior to informed consent;
2. Male and female patients on diet and exercise regimen who are drug naive, defined as absence of any oral antidiabetic therapy or insulin for 12 weeks prior to randomization
3. Glycosylated haemoglobin A1c (HbA1c) >/= 7.0% (53 mmol/mol) to </= 10.0% (86 mmol/mol) at visit 1 (screening);
4. Age>/=18 and </=80 years at visit 1(screening);
5. Body Mass Index (BMI)</= 45kg/m2 at visit 1 (screening);
6. Signed and dated written informed consent by date of visit 1 in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

1. Uncontrolled hyperglycaemia with a glucose level >240 mg/dl (13.3mmol/L) after an overnight fast during screening/placebo run-in and confirmed by a second measurement (Not on the same day);
2. Treatment with any oral antidiabetic drug or insulin within 12 weeks prior to randomization
3. Acute coronary syndrome (non-STEMI, STEMI and unstable angina pectoris),stroke or Transient ischemia attack (TIA) within 3 months prior to informed consent;
4. Indication of liver disease/Impaired hepatic function, defined by serum levels of either Aspartate aminotransferase (ALT or SGPT), alanine aminotransferase (AST or SGOT), or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined at visit 1 and/or run-in phase,
5. Impaired renal function, defined as eGFR< 60ml/min (moderate or severe renal impairment, modification of diet in renal disease (MDRD) formula) as determined during screening or at run-in phase
6. Bariatric surgery within the past two years and other gastrointestinal surgeries that induced chronic malabsorption
7. Medical history of Cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years
8. Blood dyscrasia or any other disorders causing haemolysis or unstable Red Blood Cell (eg. malaria, babesiosis, haemolytic anemia)
9. Known history of pancreatitis and chronic pancreatitis
10. Contraindications to metformin according to the local label
11. Treatment with anti-obesity drugs 3 months prior to informed consent or any other treatment at the time of screening (i.e. surgery, aggressive diet regimen etc) leading to unstable body weight
12. Current treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent or any other uncontrolled endocrine disorder except T2DM
13. Pre-menopausal women (last menstruation less than 1 year prior to informed consent) who:

    1. are nursing or pregnant or
    2. are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial or who do not agree to continue contraception for at least 30 days after the last dose of study drug. Acceptable methods of birth control include tubal ligation, transdermal patch, intra-uterine devices/systems(IUDs/IUSs), oral, implantable, or injectable contraceptives, complete sexual abstinence (if acceptable by local authorities), double barrier method and vasectomized partner.
14. Alcohol or drug abuse within 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake
15. Participation in another trial with application of any investigational drug within 30 days prior to informed consent
16. Any other clinical condition that would jeopardize patients safety while participating in this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (90):
- Bangladesh (3):
  - 1218.60.90001 Boehringer Ingelheim Investigational Site, Dhaka
  - 1218.60.90002 Boehringer Ingelheim Investigational Site, Dhaka
  - 1218.60.90003 Boehringer Ingelheim Investigational Site, Dhaka
- Belgium (5):
  - 1218.60.32001 Boehringer Ingelheim Investigational Site, Genk
  - 1218.60.32005 Boehringer Ingelheim Investigational Site, Ham
  - 1218.60.32002 Boehringer Ingelheim Investigational Site, Hasselt
  - 1218.60.32004 Boehringer Ingelheim Investigational Site, Natoye
  - 1218.60.32003 Boehringer Ingelheim Investigational Site, Tremelo
- Canada (15):
  - 1218.60.20009 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1218.60.20003 Boehringer Ingelheim Investigational Site, Burnaby, British Columbia
  - 1218.60.20014 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 1218.60.20010 Boehringer Ingelheim Investigational Site, Surrey, British Columbia
  - 1218.60.20004 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1218.60.20012 Boehringer Ingelheim Investigational Site, Corunna, Ontario
  - 1218.60.20015 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1218.60.20006 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1218.60.20013 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1218.60.20002 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1218.60.20011 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1218.60.20005 Boehringer Ingelheim Investigational Site, Strathroy, Ontario
  - 1218.60.20007 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1218.60.20016 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1218.60.20001 Boehringer Ingelheim Investigational Site, Saint Romuald, Quebec
- China (12):
  - 1218.60.86001 Boehringer Ingelheim Investigational Site, Beijing
  - 1218.60.86003 Boehringer Ingelheim Investigational Site, Beijing
  - 1218.60.86011 Boehringer Ingelheim Investigational Site, Changsha
  - 1218.60.86012 Boehringer Ingelheim Investigational Site, Chengdu
  - 1218.60.86010 Boehringer Ingelheim Investigational Site, Chongqing
  - 1218.60.86013 Boehringer Ingelheim Investigational Site, Hubei
  - 1218.60.86014 Boehringer Ingelheim Investigational Site, Hubei
  - 1218.60.86006 Boehringer Ingelheim Investigational Site, Nanjing
  - 1218.60.86007 Boehringer Ingelheim Investigational Site, Nanjing
  - 1218.60.86005 Boehringer Ingelheim Investigational Site, Shanghai
  - 1218.60.86009 Boehringer Ingelheim Investigational Site, Shenyang
  - 1218.60.86008 Boehringer Ingelheim Investigational Site, Wuxi
- Germany (8):
  - 1218.60.49007 Boehringer Ingelheim Investigational Site, Berlin
  - 1218.60.49008 Boehringer Ingelheim Investigational Site, Berlin
  - 1218.60.49005 Boehringer Ingelheim Investigational Site, Dresden
  - 1218.60.49004 Boehringer Ingelheim Investigational Site, Erfurt
  - 1218.60.49006 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1218.60.49003 Boehringer Ingelheim Investigational Site, Hamburg
  - 1218.60.49002 Boehringer Ingelheim Investigational Site, Neuwied
  - 1218.60.49001 Boehringer Ingelheim Investigational Site, Unterschneidheim
- Guatemala (3):
  - 1218.60.50001 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1218.60.50002 Boehringer Ingelheim Investigational Site, Guatemala City
  - 1218.60.50003 Boehringer Ingelheim Investigational Site, Guatemala City
- Hong Kong (2):
  - 1218.60.85001 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1218.60.85002 Boehringer Ingelheim Investigational Site, Hong Kong
- India (8):
  - 1218.60.91004 Boehringer Ingelheim Investigational Site, Aurangabad
  - 1218.60.91010 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.60.91005 Boehringer Ingelheim Investigational Site, Coimbatore
  - 1218.60.91008 Boehringer Ingelheim Investigational Site, Kolkata
  - 1218.60.91001 Boehringer Ingelheim Investigational Site, Nagpur
  - 1218.60.91007 Boehringer Ingelheim Investigational Site, Nagpur
  - 1218.60.91003 Boehringer Ingelheim Investigational Site, Pune
  - 1218.60.91006 Boehringer Ingelheim Investigational Site, Pune
- Lebanon (5):
  - 1218.60.96001 Boehringer Ingelheim Investigational Site, Beirut
  - 1218.60.96002 Boehringer Ingelheim Investigational Site, Beirut
  - 1218.60.96004 Boehringer Ingelheim Investigational Site, Byblos
  - 1218.60.96003 Boehringer Ingelheim Investigational Site, Hazmiyeh
  - 1218.60.96005 Boehringer Ingelheim Investigational Site, Saida
- Mexico (5):
  - 1218.60.52005 Boehringer Ingelheim Investigational Site, Aguascalientes
  - 1218.60.52003 Boehringer Ingelheim Investigational Site, Cuernavaca
  - 1218.60.52001 Boehringer Ingelheim Investigational Site, Durango
  - 1218.60.52002 Boehringer Ingelheim Investigational Site, Durango
  - 1218.60.52004 Boehringer Ingelheim Investigational Site, Monterrey
- Peru (3):
  - 1218.60.51001 Boehringer Ingelheim Investigational Site, Lima
  - 1218.60.51002 Boehringer Ingelheim Investigational Site, Lima
  - 1218.60.51004 Boehringer Ingelheim Investigational Site, Piura
- Philippines (5):
  - 1218.60.63001 Boehringer Ingelheim Investigational Site, Cebu City, Philippines
  - 1218.60.63004 Boehringer Ingelheim Investigational Site, Iloilo City, Philippines
  - 1218.60.63003 Boehringer Ingelheim Investigational Site, Manila
  - 1218.60.63002 Boehringer Ingelheim Investigational Site, Marikina City, Philippines
  - 1218.60.63005 Boehringer Ingelheim Investigational Site, Quezon City
- Spain (10):
  - 1218.60.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 1218.60.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1218.60.34003 Boehringer Ingelheim Investigational Site, Barcelona
  - 1218.60.34004 Boehringer Ingelheim Investigational Site, Barcelona
  - 1218.60.34006 Boehringer Ingelheim Investigational Site, Borges Del Camp- Tarragona
  - 1218.60.34005 Boehringer Ingelheim Investigational Site, Centelles
  - 1218.60.34009 Boehringer Ingelheim Investigational Site, Granada
  - 1218.60.34008 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1218.60.34007 Boehringer Ingelheim Investigational Site, Mataró
  - 1218.60.34010 Boehringer Ingelheim Investigational Site, Valencia
- Taiwan (6):
  - 1218.60.88006 Boehringer Ingelheim Investigational Site, Chiayi County
  - 1218.60.88003 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1218.60.88001 Boehringer Ingelheim Investigational Site, Taichung
  - 1218.60.88007 Boehringer Ingelheim Investigational Site, Taichung
  - 1218.60.88002 Boehringer Ingelheim Investigational Site, Tainan
  - 1218.60.88004 Boehringer Ingelheim Investigational Site, Taipei County

REFERENCES:
- [Derived] Ji L, Zinman B, Patel S, Ji J, Bailes Z, Thiemann S, Seck T. Efficacy and safety of linagliptin co-administered with low-dose metformin once daily versus high-dose metformin twice daily in treatment-naive patients with type 2 diabetes: a double-blind randomized trial. Adv Ther. 2015 Mar;32(3):201-15. doi: 10.1007/s12325-015-0195-3. Epub 2015 Mar 25. PMID 25805187

RESULTS

PARTICIPANT FLOW:
Groups:
- Lina 5mg + Met qd: Patients treated with Linagliptin 5mg in combination with metformin once daily.
- Met Bid: Patients treated with metformin alone twice daily.
Period: Overall Study
Arm/Group | Lina 5mg + Met qd | Met Bid
Started | 344 | 345
Completed | 330 | 331
Not Completed | 14 | 14
Not completed — Adverse Event | 3 | 3
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Other | 2 | 4

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all patients treated with at least 1 dose of randomised study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Lina 5mg + Met qd | Met Bid | Total
Number analyzed (Participants) | 344 | 345 | 689
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (10.7) | 52.9 (10.7) | 53.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 187 | 362
  Male | 169 | 158 | 327

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin A1c (HbA1c) After 14 Weeks Treatment
Description: Adjusted mean change in HbA1c from baseline at Week 14 was analysed using an ANCOVA model. The Model included treatment and continuous baseline HbA1c.
Time Frame: Baseline and 14 weeks
Population: FAS1000mg with last observation carried forward (LOCF): all patients randomised and treated who had a baseline at least 1 on-treatment HbA1c value and who tolerated a daily metformin dose of at least 1000 mg at the end of the titration phase.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Lina 5mg + Met qd | Met Bid
Number analyzed (Participants) | 298 | 341
percent | -0.99 (0.05) | -0.98 (0.04)
Statistical Analysis 1: Comparison: Lina 5mg + Met qd vs Met Bid; Test type: Non-Inferiority or Equivalence — One-sided test relative to 0.35; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.13 to 0.12], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Lina 5mg + Met qd vs Met Bid; Test type: Superiority or Other; p = 0.8924, ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI [-0.13 to 0.12], Standard Error of Mean 0.06

2. Secondary Outcome: Composite Endpoint of Occurrence of Treat to Target Efficacy Response, That is an HbA1c Under Treatment of <7.0% After 14 Weeks of Treatment, on no Occurrence of Moderate or Severe Gastrointestinal (GI) Side Effects During 14 Weeks of Treatment
Description: The proportion of patients who achieved all the targets in a composite endpoint (HbA1c below 7.0% after 14 weeks of treatment; no occurrence of pre-specified moderate or severe gastrointestinal (GI) side effects of metformin, as assessed by the investigators during 14 weeks of treatment)
Time Frame: 14 weeks
Population: Patients from FAS1000 with non-completer considered as failure (NCF) having a baseline HbA1c>=7.0%.
Measure: Number; unit: participants
Arm/Group | Lina 5mg + Met qd | Met Bid
Number analyzed (Participants) | 257 | 306
participants | 119 | 148
Statistical Analysis 1: Comparison: Lina 5mg + Met qd vs Met Bid; Test type: Superiority or Other; p = 0.8201, Regression, Logistic; Model includes treatment and continuous baseline HbA1c; Odds Ratio (OR) = 0.960, 95% CI [0.672 to 1.370]

3. Secondary Outcome: Occurence of Metformin Pre-specified Moderate to Severe GI Side Effects Assessed by Investigators During 14 Weeks of Treatment
Description: Proportion of patients who experienced at least one metformin pre-specified moderate or severe GI side effect during 14 weeks
Time Frame: 14 weeks
Population: Patients from FAS1000
Measure: Number; unit: participants
Arm/Group | Lina 5mg + Met qd | Met Bid
Number analyzed (Participants) | 298 | 341
participants | 25 | 28
Statistical Analysis 1: Comparison: Lina 5mg + Met qd vs Met Bid; Test type: Superiority or Other; p = 0.9397, Regression, Logistic; Model includes treatment and baseline HbA1c; Odds Ratio (OR) = 1.022, 95% CI 2-sided [0.582 to 1.796]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 14 Weeks of Treatment
Description: Means are adjusted by treatment, continuous baseline HbA1c and continuous baseline fasting plasma glucose.
Time Frame: Baseline and 14 weeks
Population: Patients from FAS1000 with LOCF
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Lina 5mg + Met qd | Met Bid
Number analyzed (Participants) | 298 | 338
mg/dL | -24.5 (1.5) | -26.6 (1.4)
Statistical Analysis 1: Comparison: Lina 5mg + Met qd vs Met Bid; Test type: Superiority or Other; p = 0.3352, ANCOVA; Mean Difference (Final Values) = 2.0, 95% CI [-2.1 to 6.1], Standard Error of Mean 2.1

5. Secondary Outcome: Metformin Pre-specified GI Symptom Intensity Score Assessed by Investigators During 14 Weeks of Treatment
Description: Patients could experience multiple events, therefore, multiple answers were possible for each patient.
Time Frame: 14 weeks
Population: Patients from FAS1000 and having GI adverse events which were assessed for severity by the investigator.
Measure: Number; unit: events
Units Other Than Participants: Events
Arm/Group | Lina 5mg + Met qd | Met Bid
Number analyzed (Participants) | 73 | 98
Number analyzed (Events) | 157 | 219
events
  Mild | 114 | 153
  Moderate | 37 | 65
  Severe | 6 | 1
Statistical Analysis 1: Comparison: Lina 5mg + Met qd vs Met Bid; Test type: Superiority or Other; p = 0.0308, Fisher Exact; Fishers exact p-value presented due to small cell counts

6. Secondary Outcome: Metformin Pre-specified GI Symptom Intensity Score Assessed by Patients During 14 Weeks of Treatment
Description: The intensity of the GI side effects was also assessed by the patients using VAS scaled from 0 to 10; higher scores indicate more severe events. Means are adjusted by treatment and continuous baseline HbA1c.
Time Frame: 14 weeks
Population: Patients from the FAS1000 using original results (OR) and having GI adverse events which were assessed for severity by the patient.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lina 5mg + Met qd | Met Bid
Number analyzed (Participants) | 154 | 209
units on a scale | 4.9 (0.2) | 4.4 (0.2)
Statistical Analysis 1: Comparison: Lina 5mg + Met qd vs Met Bid; Test type: Superiority or Other; p = 0.0545, ANCOVA; Mean Difference (Final Values) = 0.5, 95% CI [-0.0 to 1.0], Standard Error of Mean 0.3

7. Secondary Outcome: Composite Endpoint of Occurrence of Treat to Target Efficacy Response, That is an HbA1c Under Treatment of <6.5% After 14 Weeks of Treatment, and no Occurrence of Moderate or Severe Metformin Pre-specified GI Side Effects Assessed by Investigators
Description: The proportion of patients who achieved all the targets in a composite endpoint (HbA1c below 6.5% after 14 weeks of treatment; no occurrence of pre-specified moderate or severe GI side effects of metformin, as assessed by the investigators during 14 weeks of treatment).
Time Frame: 14 weeks
Population: Patients from FAS1000 (NCF) having a baseline HbA1c>=6.5%.
Measure: Number; unit: participants
Arm/Group | Lina 5mg + Met qd | Met Bid
Number analyzed (Participants) | 291 | 338
participants | 83 | 95
Statistical Analysis 1: Comparison: Lina 5mg + Met qd vs Met Bid; Test type: Superiority or Other; p = 0.9886, Regression, Logistic; Odds Ratio (OR) = 0.997, 95% CI [0.689 to 1.445]

8. Secondary Outcome: Occurrence of Relative Efficacy Response (HbA1c Lowering by at Least 0.5% After 14 Weeks of Treatment)
Description: The proportion of patients who achieved a relative efficacy response (HbA1c lowering by at least 0.5% after 14 weeks of treatment).
Time Frame: 14 weeks
Population: Patients from FAS1000 (NCF)
Measure: Number; unit: participants
Arm/Group | Lina 5mg + Met qd | Met Bid
Number analyzed (Participants) | 298 | 341
participants | 211 | 257
Statistical Analysis 1: Comparison: Lina 5mg + Met qd vs Met Bid; Test type: Superiority or Other; p = 0.2108, Regression, Logistic; Odds Ratio (OR) = 0.797, 95% CI [0.558 to 1.137]

9. Secondary Outcome: Occurrence of Relative Efficacy Response (HbA1c Lowering by at Least 0.8% After 14 Weeks of Treatment)
Description: The proportion of patients who achieved a relative efficacy response (HbA1c lowering by at least 0.8% after 14 weeks of treatment).
Time Frame: 14 weeks
Population: Patients from the FAS1000 (NCF)
Measure: Number; unit: participants
Arm/Group | Lina 5mg + Met qd | Met Bid
Number analyzed (Participants) | 298 | 341
participants | 162 | 187
Statistical Analysis 1: Comparison: Lina 5mg + Met qd vs Met Bid; Test type: Superiority or Other; p = 0.9972, Regression, Logistic; Odds Ratio (OR) = 0.999, 95% CI [0.712 to 1.402]

10. Secondary Outcome: Composite Endpoint of Occurence of Relative Efficacy Response (HbA1c Lowering by at Least 0.5% After 14 Weeks of Treatment) and no Occurence of Moderate and Severe Metformin Pre-specified GI Side Effects Assessed by the Investigators During 14 Weeks
Description: The proportion of patients who achieved all the targets in a composite endpoint (HbA1c lowered by at least 0.5% after 14 weeks of treatment; no occurrence of pre-specified moderate or severe GI side effects of metformin, as assessed by the investigators during 14 weeks of treatment).
Time Frame: 14 weeks
Population: Patients from FAS1000 (NCF)
Measure: Number; unit: participants
Arm/Group | Lina 5mg + Met qd | Met Bid
Number analyzed (Participants) | 298 | 341
participants | 194 | 236
Statistical Analysis 1: Comparison: Lina 5mg + Met qd vs Met Bid; Test type: Superiority or Other; p = 0.2816, Regression, Logistic; Odds Ratio (OR) = 0.832, 95% CI [0.594 to 1.163]

11. Secondary Outcome: Change From Baseline in Body Weight by Visit at Week 14
Description: Means are adjusted by treatment, continuous baseline HbA1c and continuous baseline weight
Time Frame: Baseline and 14 weeks
Population: FAS1000 having values for weight at baseline and week 14.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Lina 5mg + Met qd | Met Bid
Number analyzed (Participants) | 287 | 324
kg | -0.44 (0.14) | -1.05 (0.13)
Statistical Analysis 1: Comparison: Lina 5mg + Met qd vs Met Bid; Test type: Superiority or Other; p = 0.0011, ANCOVA; Mean Difference (Final Values) = 0.62, 95% CI [0.25 to 0.98], Standard Error of Mean 0.19

12. Secondary Outcome: Composite Endpoint of Occurrence of Relative Efficacy Response (HbA1c Lowering by at Least 0.8% After 14 Weeks of Treatment) and no Occurrence of Moderate and Severe Metformin Pre-specified GI Side Effects Assessed by Investigators During 14 Weeks
Description: The proportion of patients who achieved all the targets in a composite endpoint (HbA1c lowered by at least 0.8% after 14 weeks of treatment; no occurrence of pre-specified moderate or severe GI side effects of metformin, as assessed by the investigators during 14 weeks of treatment).
Time Frame: 14 weeks
Population: Patients from FAS1000 (NCF)
Measure: Number; unit: participants
Arm/Group | Lina 5mg + Met qd | Met Bid
Number analyzed (Participants) | 298 | 341
participants | 149 | 175
Statistical Analysis 1: Comparison: Lina 5mg + Met qd vs Met Bid; Test type: Superiority or Other; p = 0.7682, Regression, Logistic; Odds Ratio (OR) = 0.951, 95% CI [0.681 to 1.328]

13. Secondary Outcome: Change From Baseline in HbA1c Over Time
Description: Means are adjusted by treatment and continuous baseline HbA1c
Time Frame: Baseline, 2 weeks and 8 weeks
Population: Patients from FAS1000 (LOCF)
Measure: Mean (Standard Error); unit: percent
Arm/Group | Lina 5mg + Met qd | Met Bid
Number analyzed (Participants) | 298 | 341
percent
  At week 2 | -0.28 (0.02) | -0.25 (0.02)
  At week 8 | -0.84 (0.04) | -0.78 (0.04)

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Lina 5mg + Met qd | Met Bid
Serious Adverse Events (participants affected / at risk) | 2/344 | 7/345
Other Adverse Events (participants affected / at risk) | 101/344 | 121/345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lina 5mg + Met qd (N=344) | Met Bid (N=345)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Epiploic appendagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lina 5mg + Met qd (N=344) | Met Bid (N=345)
Abdominal pain (Gastrointestinal disorders) | 23 | 29
Diarrhoea (Gastrointestinal disorders) | 62 | 74
Nausea (Gastrointestinal disorders) | 23 | 24
Urinary tract infection (Infections and infestations) | 17 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.